CLINICAL TRIAL: NCT05505812
Title: Study on the Safety and Efficacy of Autogenous Tumor Infiltrates Lymphocytes (HS-IT101) for the Treatment of Advanced Breast Cancer
Brief Title: Study on the Safety and Efficacy of Autogenous Tumor Infiltrates Lymphocytes for the Treatment of Advanced Breast Cancer
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Collaborators: Qingdao Sino-Cell Biomedicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: wanghaibo
Record Dates: First submitted 2022-08-16; First posted 2022-08-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HS-IT101 monotherapy (Experimental): 1x10^9-6x10^10 in vitro expanded autologous TIL (HS-IT101) will be infused i.v. to patients with advanced breast cancer after lymphodepletion treatment with fludarabine and cyclophosphamide, and then followed by the administration of a regimen of IL-2.
  Interventions: Biological: HS-IT101

INTERVENTIONS:
Biological: HS-IT101 — Adoptive transfer of 1x10^9-6x10^10 autologous TIL to patients i.v. in 30-60 minutes.

SUMMARY:
Prospective, single-center, single-arm, open-label,interventional study evaluating adoptive cell therapy (ACT) with autologous tumor-infiltrating lymphocyte (TIL) infusion (HS-IT101) after lymphodepletion preparative with fludarabine and cyclophosphamide regimen, followed by IL-2, for the treatment of patients with advanced breast cancer.

DETAILED DESCRIPTION:
HS-IT101 is an adoptive cell transfer therapy that utilizes an autologous TIL manufacturing process, for the treatment of patients with advanced breast cancer. The cell transfer therapy used in this study involves patients receiving lymphodepletion treatment with fludarabine and cyclophosphamide, followed by infusion of autologous TIL, then finnaly followed by the administration of a regimen of IL-2.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for the study, patients must meet ALL of the following criteria prior to participation:

  1. Age: 18 years to 75 years at the time of consent (Female);
  2. Histologically or cytological diagnosed as advanced breast cancer;
  3. Test subjects have failed first-line standard treatment regimens, and there are no available effective treatment regimens option or refuses to accept further treatment;
  4. At least one resectable lesion that has not received radiotherapy or other local therapy within 28 days, and of aminimum 1cm∧3 resection；or resectable lesions capable of producing sufficient TIL；
  5. At least one measurable target lesion, as defined by RECIST v1.1，that has not received radiotherapy or other local therapy unless these therapies occurred 28 days ago and target lesion shows significant progression;
  6. ECOG score 0-2;
  7. Expected life-span more than 3 months;
  8. Adequate organ and bone marrow function:

     * Absolute count of neutrophil ≥1.5×10^9/L; Platelet count ≥90×10^9/L; Hemoglobin ≥ 90g/L (None blood transfusion or erythropoietin treatment within 14 days);
     * AST, ALT≤2.5×ULN (subjects with liver metastasis ≤5×ULN); Totol bilirubin ≤1.5×ULN;
     * Serum creatinine ≤1.5×ULN, or estimated creatinine clearance (CrCl)≥45 mL/min (Cockcroft-Gault formula);
     * Activated partial thromboplastin time (APTT) ≤1.5×ULN, while international no○rmalized ratio (INR) or prothrombin (PT) ≤1.5×ULN;
     * LVEF ≥ 50%, none symptomatic or poorly controlled arrhythmias;
  9. Test subjects must have recovered from all prior therapy-related toxicities to ≤Grade 1 according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0; except for alopecia (tumor resection);
  10. Test subjects with child-bearing potential must be willing to practice approved highly effective methods of contraception at the time of informed consent, and continue within 180 days after the completion of treatment；
  11. Be able to understand and sign the informed consent document.

Exclusion Criteria:

* Patients with any of the following criteria will not be allowed to participation:

  1. Test subjects who have a history of hypersensitivity to any component or excipient of HS-IT101 or other study drugs (cyclophosphamide, fludarabine and recombinant human interleukin-2);
  2. Test subjects have any uncontrollable clinical problems (including but not limited):

     * hypertension poorly controlled by medication (blood pressure ≥150/90mmHg at rest after taking medication);
     * poorly controlled diabetes;
     * cardiac disease (New York Heart Association class Ⅲ/Ⅳ congestive heart failure or heart block);
  3. Test subjects who have active major medical illnesse(es) of the cardiovascular (within 6 months prior to enrollment), including deep vein thrombosis or pulmonary embolism; myocardial infarction; severe or unstable arrhythmia or angina pectoris; percutaneous coronary intervention, acute coronary syndrome, coronary artery bypass grafting; cerebrovascular accident, transient cerebral ischemia Seizures, cerebral embolism;
  4. Active autoimmune diseases or recipients of organ transplants that require systemic treatment during the study period, or a history of such diseases within the past 2 years;
  5. Prior used any immunosuppressive medications, such as corticosteroids (within 14 days prior to enrollment); physiological doses of glucocorticoids (≤10 mg/day prednisone or equivalent) are permitted, as well as inhaled, intranasal, or topical corticosteroids;
  6. Test subjects with symptomatic and/or untreated brain metastases;
  7. Current or prior use of anticancer therapy: a.) chemotherapy, immune checkpoint inhibitor, other investigational therapy drug or local treatment for target lesions within the past 4 weeks; b.) chinese patent medicine with anti-tumor indications, or systemic therapy with immunomodulatory drugs (including thymosin, interferon, drugs targeting) within the past 2 weeks; c.) targeted drug therapy within the past 4 weeks or 5 half-lives, whichever is shorter;
  8. Presence of acute or chronic infection:

     * Human immunodeficiency virus (HIV) infection or anti-HIV antibody positive;
     * Active TB infection;
     * Active bacterial or fungal infection requiring systemic treatment;
     * HBsAg and/or HBeAg positive;
     * Hepatitis C patients;
     * Treponema pallidum antibodies positive;
  9. Vaccinated with the new coronavirus vaccine within 14 days propr to screening, or who have received a live vaccine within 3 months, or who plan to receive live vaccine during the trial;
  10. Major organs underwent surgery (excluding needle biopsy) or significant trauma within 4 weeks before screening；required elective surgery during the study;
  11. Test subjects who have had another primary malignancy within the previous 5 years, excluding basal cell carcinoma of the skin, squamous cell carcinoma of the skin and/or carcinoma in situ after radical resection;
  12. Females in pregnancy or lactation;
  13. Test subjects have had SAE requiring blood product support occurred in previous chemotherapy, including but not limited to whole blood, red blood cells, platelets;
  14. Subject have mental illness, alcoholism, drug or substance abuse；or researchers considering the test subject as having other reasons inappropriate for the clinical study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-10-08 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AE) | 12 months
  To characterize the safety profile of HS-IT101 in patients with advanced breast cancer as assessed by incidence of adverse events.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 36 months
  To evaluate the efficacy of HS-IT101 in patients with advanced breast cancer, based on the objective response rate (ORR) as assessed by the Independent Review Committee (IRC) per RECIST v1.1
Time-to-response (TTR) | Up to 36 months
  To evaluate the efficacy of HS-IT101 in patients with advanced breast cancer by assessing the time-to-response (TTR) as assessed by the Investigator per RECIST v1.1
Duration of Response (DOR) | Up to 36 months
  To evaluate the efficacy of HS-IT101 in patients with advanced breast cancer by assessing the duration of response (DOR) as assessed by the Investigator per RECIST v1.1
Overall Survival (OS) | Up to 36 months
  To evaluate overall survival (OS) in patients with advanced breast cancer

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Wang, MD, Principal Investigator — The Affiliated Hospital of Qingdao University
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No